CLINICAL TRIAL: NCT01372189
Title: In Vivo Molecular Imaging of Epidermal Growth Factor Receptor in Patients With Colorectal Neoplasia Using Confocal Laser Endomicroscopy
Brief Title: Molecular Imaging of Epidermal Growth Factor Receptor in Colorectal Neoplasia Using Confocal Laser Endomicroscopy
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Chief of the Department of Gastroenterology, Qilu Hospital, Shandong University, Shandong University
Other Study IDs: 2011SDU-QILU-G01
Record Dates: First submitted 2011-01-18; First posted 2011-06-13 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Colorectal Cancer; Colorectal Adenoma
Keywords: molecular imaging; epidermal growth factor receptor; colorectal neoplasia; confocal laser endomicroscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Take biospecimen during colonoscopy.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- colorectal cancer: Patients with colorectal carcinoma during conventional endoscopic imaging.
- colorectal adenoma: Patients with colorectal adenoma during conventional endoscopic imaging.

SUMMARY:
The study aims to:

1. Achieve molecular imaging of EGFR in patients with colorectal neoplasia in vivo using confocal laser endomicroscopy.
2. Compare the results of in vivo EGFR-specific molecular imaging with CLE and ex vivo immunohistochemistry .

DETAILED DESCRIPTION:
Various kinds of tumor markers have been shown to be over-expressed in colorectal cancer, including epidermal growth factor receptor(EGFR). The conventional detection method of EGFR expression in colorectal neoplasia is immunohistochemistry which is time-consuming, and the immunoreactivity can be affected by storage and fixation of tissues. Confocal laser endomicrosopy is a newly developed device which could identify the cellular and subcellular structures clearly with the magnification at×1000, making it possible to explore the physiological and pathological molecular mechanism of the gastrointestinal tract. So the study aims to achieve molecular imaging of EGFR in colorectal neoplasia in vivo using confocal laser endomicroscopy.

ELIGIBILITY:
Inclusion Criteria：

●Patients known to have large polypoid lesions in colon or rectum from previous examinations from outpatients and inpatients at Qilu Hospital were enrolled into the study

Exclusion Criteria:

* Patients who are allergic to fluorescein sodium
* Patients with impaired cardiac, liver or renal function
* Patients who are unwilling to sign or give the informed consent form
* Patients with giant tumors or obvious GI tract bleeding which make it hard or impossible to observe the lesions
* Patients with coagulopathy
* Patients with pregnancy or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients known to have large polypoid lesions in colon or rectum from previous examinations from outpatients and inpatients at Qilu Hospital were enrolled into the study
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD. MD., Study Director — Department of Gastroenterology, Qilu Hospital
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China